CLINICAL TRIAL: NCT01495793
Title: A Multicenter, Open-Label, 2-Group, Dose Escalation Study of Monotherapy Administration of Rotigotine in Pediatric Subjects With Idiopathic Restless Legs Syndrome
Brief Title: Dose Escalating Study of Rotigotine in Pediatric Subjects With Restless Legs Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SP1004; 2014-004383-37 (EudraCT Number)
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Results first posted 2015-07-14 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Restless Legs Syndrome
Keywords: Rotigotine; Restless Legs Syndrome; RLS; Children; Adolescents
MeSH Terms: conditions — Restless Legs Syndrome | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rotigotine (Experimental): In the Titration Period a subject received the first dose of rotigotine then the dose was increased weekly by a dose step over 4 weeks.
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — Rotigotine transdermal patch:
  Dose (size): 0.5 mg/24 h (2.5 cm^2)- 1 mg/24 h (5 cm^2)- 2 mg/24 h (10 cm^2)- 3 mg/24 h (15 cm^2) The patch has to be applied continuously for 24h. After 24h, the patch has to be removed and a new one applied.

SUMMARY:
This was a multicenter, open-label, dose-escalation, Phase 2A study with multiple administrations of the rotigotine transdermal system. The study was conducted in adolescent subjects (13 to <18 years of age) with idiopathic Restless Legs Syndrome (RLS).

ELIGIBILITY:
Inclusion Criteria:

* Subject or parent/legal representative is considered reliable and capable of adhering to the protocol
* Subject is male or female, and is ≥13 and <18 years of age at Visit 2/Baseline
* Subject weighs ≥40 kg at Visit 2/Baseline
* Subject's Body Mass Index (BMI) is less than the 95th percentile for his or her age at Visit 2/Baseline
* Subject meets the diagnosis of RLS based on the proposed 2011 Revised International Restless Legs Syndrome Study Group Diagnostic Criteria
* Subject's RLS symptoms cause significant distress or impairment
* At Visit 2/Baseline, subject has a Periodic Limb Movement Index (PLMI) ≥5 during at least 1 of the 5 nights prior to Baseline as measured by the activity monitors
* At Visit 2/Baseline, subject has a score of ≥15 on the IRLS Rating Scale
* At Visit 2/Baseline, subject scores ≥4 points on the Clinical Global Impression (CGI) Item 1 assessment
* Subject receiving supplemental iron has been on a stable dose for at least 3 months prior to Visit 1/Screening Period

Exclusion Criteria:

* Previously participated in this study or received previous treatment with rotigotine
* Participated in another study of an investigational medicinal product (IMP) or a medical device within the last 3 months prior to Visit 1/Screening Period or is currently participating in another study of an IMP or a medical device
* Subject's RLS symptoms are restricted only to the ankles or knees
* RLS symptoms are due to renal insufficiency (uremia) or iron deficiency anemia
* Previous treatment with dopamine agonists within a period of 14 days prior to Visit 2/Baseline or L-dopa within 7 days prior to Visit 2/Baseline
* Failed to respond to previous dopaminergic therapy
* Any medical or psychiatric condition, which in the opinion of the investigator, would jeopardize or compromise the subject's well being or ability to participate
* Subject has a lifetime history of suicide attempt or has suicidal ideation in the past 6 months
* Evidence of an impulse control disorder (ICD)
* History or current symptoms of sleep apnea, narcolepsy, sleep attacks/sudden onset of sleep, or myoclonus epilepsy
* Concomitant diseases such as peripheral neuropathy, muscle fasciculation, painful legs and moving toes, fibromyalgia, rheumatoid arthritis, or sickle cell disease
* Serum ferritin level <15 ng/mL
* Subject has not attempted at least 1 non-pharmacological intervention for the management of RLS (eg, sleep hygiene, exercise)
* Prior history of psychotic episodes
* History of chronic alcohol or drug abuse within 12 months prior Screening Period
* Clinically relevant cardiac dysfunction and/or arrhythmias
* Hemoglobin level below the lower limit of normal
* Clinically relevant renal dysfunction (serum creatinine >1.5 mg/dL)
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin level greater than or equal to 2 times the upper limit of normal
* History or presence of clinical signs of any malignant neoplasm including suspicious undiagnosed skin lesion (which may be melanoma), melanoma, or a history of melanoma
* Currently receiving or has received treatment with any of the following within 28 days prior to Visit 2/Baseline: neuroleptics, antidepressants, anxiolytic drugs, opioids, monoamine oxidase (MAO) inhibitors, or sedative antihistamines
* Currently receiving treatment with any of the following: benzodiazepines, hypnotics, anticonvulsants, central alpha-adrenergic agonists, or melatonin; unless treatment is for RLS only, in which case a Wash-Out Period of at least 14 days prior to Visit 2/Baseline is required
* Currently receiving stimulant therapy for attention deficit hyperactivity disorder (ADHD); a Wash-Out Period of at least 7 days prior to Visit 2/Baseline is required
* Pregnant, nursing, or is a woman of childbearing potential who is not surgically sterile, or does not consistently use 2 combined medically acceptable methods of contraception (including at least 1 barrier method), unless not sexually active
* Unwilling to abstain from caffeine after 4pm each evening within 7 days prior to Visit 2/Baseline and for the duration of the study
* Pursues shift work or performs other continuous non-disease-related life conditions, which do not allow regular sleep at night
* Subject has a QT correction (QTc) interval of ≥500 ms at Visit 1/Screening Period or Visit 2/Baseline. Bazett's correction method must be used for the correction of the QT interval
* Symptomatic orthostatic hypotension with a decrease of blood pressure (BP) from supine to standing position of ≥20 mmHg in systolic blood pressure (SBP) or of ≥10 mmHg in diastolic blood pressure (DBP) taken from the 5 minute supine and 1 and/or 3 minute standing measurements
* A known hypersensitivity to any of the components of the study medication, such as a history of significant skin hypersensitivity to adhesives, known hypersensitive

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2011-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — 1-877-822-9493 (UCB)
Locations (12):
- United States (12):
  - Sp1004 006, Little Rock, Arkansas
  - Sp1004 012, Los Angeles, California
  - Sp1004 009, Orange, California
  - Sp1004 005, Washington D.C., District of Columbia
  - Sp1004 014, Spring Hill, Florida
  - Sp1004 013, Indianapolis, Indiana
  - Sp1004 001, Destrehan, Louisiana
  - Sp1004 015, St Louis, Missouri
  - Sp1004 007, West Seneca, New York
  - Sp1004 002, Cincinnati, Ohio
  - Sp1004 016, West Chester, Pennsylvania
  - Sp1004 003, Austin, Texas

REFERENCES:
- [Result] Elshoff JP, Hudson J, Picchietti DL, Ridel K, Walters AS, Doggett K, Moran K, Oortgiesen M, Ramirez F, Schollmayer E. Pharmacokinetics of rotigotine transdermal system in adolescents with idiopathic restless legs syndrome (Willis-Ekbom disease). Sleep Med. 2017 Apr;32:48-55. doi: 10.1016/j.sleep.2016.04.012. Epub 2016 Jun 8. PMID 28366342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study in which 42 subjects were enrolled and 24 treated at 8 sites in the USA.
Pre-assignment Details: In total 42 subjects signed the informed consent and were enrolled into the study (Enrolled Set). 24 of these subjects were treated with medication. The sample size of 24 subjects was sufficient to target a 95% confidence interval and the calculation was based on a previous study. Participant Flow refers to the 24 treated subjects (Safety Set).
Period: Overall Study
Arm/Group | Rotigotine
Started | 24
Completed | 22
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Violation of inclusion criteria | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refers to the 24 treated subjects (Safety Set).
Arm/Group | Rotigotine
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (1.3)
Age, Customized [Number; unit: Participants]
  13 years | 2
  14 years | 6
  15 years | 6
  16 years | 4
  17 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: cm] | 167.39 (6.89)
Weight [Mean (Standard Deviation); unit: kg] | 65.70 (10.72)
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] | 23.388 (3.133)

OUTCOME MEASURES:

1. Primary Outcome: Apparent Total Body Clearance (Cl/f) of Unconjugated Rotigotine 0.5 mg/24 h (2.5 cm^2)
Description: CL/f was calculated for each subject treated with rotigotine derived from the concentrations of unconjugated rotigotine measured in plasma.
  For the primary variables the parametric point estimator for each dose step and the 95% CI was calculated using the least-squares (LS) means and the root mean square of error from the ANOVA of the log-transformed data with subsequent exponential transformation.
Time Frame: 0 h (predose), 1 h, 2 h, 7-12 h and 22-24 h on Day 7, 14, 21 and 28
Population: The Pharmacokinetic Per Protocol Set (PKPPS) includes all enrolled subjects who were included in the Safety Set, who had no protocol deviations that were considered to impact the subject's validity for analysis of the primary study objective and who for at least 1 dose step fulfilled specific predefined conditions.
Measure: Least Squares Mean (95% Confidence Interval); unit: L/h (liter per hour)
Groups:
- Rotigotine (PKPPS): In the Titration Period a subject received the first dose of rotigotine then the dose was increased weekly by a dose step over 4 weeks.
Arm/Group | Rotigotine (PKPPS)
Number analyzed (Participants) | 6
L/h (liter per hour) | 676.86 [408.50 to 1121.51]

2. Primary Outcome: Apparent Total Body Clearance (Cl/f) of Unconjugated Rotigotine 1 mg/24 h (5 cm^2)
Description: as for outcome 1
Time Frame: 0 h (predose), 1 h, 2 h, 7-12 h and 22-24 h on Day 7, 14, 21 and 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: L/h (Liter per hour)
Arm/Group | Rotigotine (PKPPS)
Number analyzed (Participants) | 10
L/h (Liter per hour) | 671.72 [459.11 to 982.80]

3. Primary Outcome: Apparent Total Body Clearance (Cl/f) of Unconjugated Rotigotine 2 mg/24 h (10 cm^2)
Description: as for outcome 1
Time Frame: 0 h (predose), 1 h, 2 h, 7-12 h and 22-24 h on Day 7, 14, 21 and 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: L/h (Liter per hour)
Arm/Group | Rotigotine (PKPPS)
Number analyzed (Participants) | 11
L/h (Liter per hour) | 937.56 [658.50 to 1334.89]

4. Primary Outcome: Apparent Total Body Clearance (Cl/f) of Unconjugated Rotigotine 3 mg/24 h (15 cm^2)
Description: as for outcome 1
Time Frame: 0 h (predose), 1 h, 2 h, 7-12 h and 22-24 h on Day 7, 14, 21 and 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: L/h (Liter per hour)
Arm/Group | Rotigotine (PKPPS)
Number analyzed (Participants) | 9
L/h (Liter per hour) | 1088.77 [723.47 to 1638.53]

5. Primary Outcome: Volume of Distribution at Steady State (VSS/f) of Unconjugated Rotigotine 0.5 mg/24 h (2.5 cm^2)
Description: VSS/f was calculated for each subject treated with rotigotine derived from the concentrations of unconjugated rotigotine measured in plasma.
  For the primary variables the parametric point estimator for each dose step and the 95% CI was calculated using the least-squares (LS) means and the root mean square of error from the ANOVA of the log-transformed data with subsequent exponential transformation.
Time Frame: 0 h (predose), 1 h, 2 h, 7-12 h and 22-24 h on Day 7, 14, 21 and 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: L (Liter)
Arm/Group | Rotigotine (PKPPS)
Number analyzed (Participants) | 6
L (Liter) | 5403.16 [2850.67 to 10241.17]

6. Primary Outcome: Volume of Distribution at Steady State (VSS/f) of Unconjugated Rotigotine 1 mg/24 h (5 cm^2)
Description: as for outcome 5
Time Frame: 0 h (predose), 1 h, 2 h, 7-12 h and 22-24 h on Day 7, 14, 21 and 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: L (Liter)
Arm/Group | Rotigotine (PKPPS)
Number analyzed (Participants) | 10
L (Liter) | 6220.79 [3842.05 to 10072.28]

7. Primary Outcome: Volume of Distribution at Steady State (VSS/f) of Unconjugated Rotigotine 2 mg/24 h (10 cm^2)
Description: as for outcome 5
Time Frame: 0 h (predose), 1 h, 2 h, 7-12 h and 22-24 h on Day 7, 14, 21 and 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: L (Liter)
Arm/Group | Rotigotine (PKPPS)
Number analyzed (Participants) | 11
L (Liter) | 7114.01 [4547.88 to 11128.07]

8. Primary Outcome: Volume of Distribution at Steady State (VSS/f) of Unconjugated Rotigotine 3 mg/24 h (15 cm^2)
Description: as for outcome 5
Time Frame: 0 h (predose), 1 h, 2 h, 7-12 h and 22-24 h on Day 7, 14, 21 and 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: L (Liter)
Arm/Group | Rotigotine (PKPPS)
Number analyzed (Participants) | 9
L (Liter) | 6037.92 [3598.36 to 10131.41]

ADVERSE EVENTS:
Time Frame: This summary includes TEAEs from the Titration period, Taper period and Safety Follow-up (Day 1 up to 69 days).
Arm/Group | Rotigotine
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 15/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=24)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (11)
Vomiting (Gastrointestinal disorders) | 2 (2)
Application site pruritus (General disorders) | 4 (4)
Application site irritation (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 1 (1)
Food allergy (Immune system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (3)
Pharyngitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscukoseletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Migraine (Nervous system disorders) | 1 (1)
Dizzines (Nervous system disorders) | 2 (2)
Sudden onset of sleep (Nervous system disorders) | 1 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days